CLINICAL TRIAL: NCT03530072
Title: Using Next Gen Sequencing to Identify Pediatric Patients With Febrile Neutropenia at Low Risk for Complications: A Pilot Study
Brief Title: Use of NGS Cell-free Pathogen Test for Identification of Low Risk Fever & Neutropenia in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Karius, Inc. (Industry)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: KDP-005
Record Dates: First submitted 2018-05-07; First posted 2018-05-21 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Neutropenia; Fever
MeSH Terms: conditions — Neutropenia; Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases: Subjects with Fever and Neutropenia
  Interventions: Diagnostic Test: Karius Test

INTERVENTIONS:
Diagnostic Test: Karius Test — Next Generation Sequencing

SUMMARY:
Febrile neutropenia is a common complication in pediatric oncology patients. Standard of care requires admission of all patients for intravenous antibiotics until cultures are negative, patients are afebrile and there are signs of bone marrow recovery. This often results in prolonged hospital admissions with significant financial costs, decreased quality of life and potential secondary infections. More recent data suggests it may be possible to identify a "low risk" group that can be discharged prior to signs of bone marrow recovery. At this time, researchers have been unable to identify a model that is safe for early discharge across institutions.

DETAILED DESCRIPTION:
1. Conduct a pilot study to determine the feasibility of using the Karius Assay to risk stratify pediatric oncology patients admitted with febrile neutropenia. This will provide preliminary data for a larger study which would randomize patients to early discharge vs. usual care.
2. Evaluate the Klaasen and SPOG clinical decision rules with and without the Karius Assay to predict patients at low risk for adverse infectious outcomes during admission. Adverse infectious outcome will be defined as: positive blood or urine culture, radiographic evidence of infection, admission to the intensive care unit or death.
3. Model potential cost savings of early discharge for patients deemed low risk for an adverse infectious outcome.

ELIGIBILITY:
Inclusion Criteria:

1) Pediatric oncology patients, aged 1-22, treated at Lucile Packard Children's Hospital (LPCH)

Exclusion Criteria:

1. Relapsed disease
2. Acute lymphoblastic leukemia during induction
3. Acute myeloid leukemia during any phase of treatment
4. Philadelphia-chromosome positive ALL
5. Down syndrome
6. Patients who have received an allogeneic stem cell transplant.

Ages: 1 Year to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children being admitted for inpatient treatment with fever and neutropenia.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Modeled sensitivity and specificity | 1 day of Discharge
  Sensitivity, specificity, PPV, NPV of Klassen and SPOG clinical decision rules with and without incorporation of Karius test for prediction of patients at low risk for infectious outcomes during hospital admission. Assessed at time of Discharge

SECONDARY OUTCOMES:
Modeled cost savings | 1 day of Discharge
  Estimate cost savings for hospital stay with and without Karius results at time of discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Aftandillian, MD, Principal Investigator — Lucille Packard Children's Hospital/Stanford University
Locations (1):
- Lucille Packard Children's Hopsital, Stanford, California, United States